CLINICAL TRIAL: NCT05052580
Title: Test to Stay in School: COVID-19 Testing Following Exposure in School Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00109436
Record Dates: First submitted 2021-09-20; First posted 2021-09-22 (Actual); Results first posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 Exposure Testing (Other)
  Interventions: Other: COVID-19 Testing

INTERVENTIONS:
Other: COVID-19 Testing — Participants who consent to participate in this study will be tested at days 1, 3, 5, and 7 following a known COVID-19 exposure on day 0. If the COVID-19 tests are negative, the participant will remain in the school environment. A positive COVID-19 test or the development of symptoms on any day after exposure would require isolation according to school, local and state guidelines.

SUMMARY:
Participants in school communities who have been exposed to SARS-CoV-2 will be tested for COVID-19 on the day of exposure (day 1) and at days 3, 5, and 7 following initial known exposure. Mitigation practices including masking, the context of exposure (classroom, school bus, after school sporting event, lunch, etc.), and results of COVID-19 test will be documented.

DETAILED DESCRIPTION:
This is a prospective, interventional study with a primary objective of evaluating severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) transmission following exposure in Kindergarten through 12th grade schools. Participants will be tested with a COVID-19 testing kit that is Food and Drug Administration (FDA)-authorized under an emergency use authorization (EUA) for non-prescription use for both symptomatic and asymptomatic evaluation in children and adults. Participants who consent to participate in this study will be tested at days 1, 3, 5, and 7 following a known COVID-19 exposure on day 0. If a participant does not know of the exposure until more than one day following they exposure, they will be tested on the day they become aware of the exposure and then resume the aforementioned testing schedule (e.g. participant identifies exposure 3 days after the exposure, test on day 3, day 5, and day 7).

If the COVID-19 tests are negative, the participant will remain in the school environment. A positive COVID-19 test or the development of symptoms on any day after exposure would require isolation according to school, local and state guidelines. Demographic information, daily presence or absence of symptoms, whether the infected person or close contact was masked, setting of the exposure, test results, and school absences will be collected following consent. Data regarding school level mitigation practices will also be collected. Data collected from this study may be combined with school-provided data and publically available community data.

ELIGIBILITY:
Inclusion Criteria:

* Consent completed
* Child or adult that is part of a school community
* Known exposure to SARS-CoV-2 in the school setting (e.g. school bus, classroom, school sporting event, etc.)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4733 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanecia Zimmerman, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Participating NC School Districts, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Campbell MM, Benjamin DK, Mann T, Fist A, Kim H, Edwards L, Rak Z, Brookhart MA, Anstrom K, Moore Z, Tilson EC, Kalu IC, Boutzoukas AE, Moorthy GS, Uthappa D, Scott Z, Weber DJ, Shane AL, Bryant KA, Zimmerman KO; ABC SCIENCE COLLABORATIVE. Test-to-Stay After Exposure to SARS-CoV-2 in K-12 Schools. Pediatrics. 2022 May 1;149(5):e2021056045. doi: 10.1542/peds.2021-056045. PMID 35437593

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COVID-19 Exposure Testing
Started | 4733
Completed | 3489 (Analysis eligible population: participants who were tested positive or had a negative follow-up test at day 5 or later, and completed follow-up among those enrolled)
Not Completed | 1244

BASELINE CHARACTERISTICS:
Population: Participants who tested positive or had a negative follow-up test at day 5 or later, and completed follow-up among those enrolled.
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 3489
Age, Continuous [Mean (Full Range); unit: years] — Population: Age was not collected as part of this study.
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 1870
  Male | 1609
  Prefer not to say | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 383
  Not Hispanic or Latino | 3092
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 17
  Asian | 66
  Native Hawaiian or Other Pacific Islander | 9
  Black or African American | 422
  White | 2780
  More than one race | 152
  Unknown or Not Reported | 43
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3489

OUTCOME MEASURES:

1. Primary Outcome: Number of Students With Positive COVID-19 Test Following Known Within-school Exposure.
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: Student participants who were tested positive or had a negative follow-up test at day 5 or later, and completed follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 3002
Participants | 285

2. Primary Outcome: Number of Staff With Positive COVID-19 Tests Following Known Within-school Exposure.
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: Staff participants who were tested positive or had a negative follow-up test at day 5 or later, and completed follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 250
Participants | 38

3. Primary Outcome: Number of Exposed Participants (as Measured by Nurse Report) Undergoing the Test-to-stay Protocol That Result in Additional Transmission.
Description: Exposures That Result in Additional Transmission (TAR = # of positives in TTS close contacts, out of all TTS close contacts)
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: Exposed participants (as measured by nurse report) undergoing the test-to-stay protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 409
Participants | 29

4. Primary Outcome: Time (in Days) to Test Positivity (Reported as a Mean) Among Those Exposed to SARS-CoV-2 and Undergoing the Test-to-stay Protocol.
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: Positive student and staff participants.
Measure: Mean (Full Range); unit: Days
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 323
Days | 3.39 [0 to 10]

5. Secondary Outcome: Number of Masked Students Who Were Exposed From Masked Versus Unmasked Individuals.
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: Masked student participants.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 3161
Participants
  COVID-19 Positive - Masked | 10
  COVID-19 Positive - Unmasked | 5
  COVID-19 Negative | 3146

6. Secondary Outcome: Number of Masked Staff Who Were Exposed From Masked Compared to Unmasked Individuals.
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: Masked staff participants.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 356
Participants
  COVID-19 Positive - Masked | 1
  COVID-19 Positive - Unmasked | 1
  COVID-19 Negative | 354

7. Secondary Outcome: Number of Unmasked Students Who Were Exposed From Masked Compared to Unmasked Individuals.
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: Unmasked student participants.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 3161
Participants
  COVID-19 Positive - Masked | 15
  COVID-19 Positive - Unmasked | 254
  COVID-19 Negative | 2892

8. Secondary Outcome: Number of Unmasked Staff Who Were Exposed From Masked Compared to Unmasked Individuals.
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: Unmasked staff participants.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 356
Participants
  COVID-19 Positive - Masked | 0
  COVID-19 Positive - Unmasked | 54
  COVID-19 Negative | 302

9. Secondary Outcome: Number of Students With Positive COVID-19 Test After Indoor vs. Outdoor Exposure.
Description: Students With Positive COVID-19 Test After Indoor vs. Outdoor Exposure
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 3161
Participants
  COVID-19 Positive - Indoor | 305
  COVID-19 Positive - Outdoor | 0
  COVID-19 Negative | 2856

10. Secondary Outcome: Number of Students With Positive COVID-19 Test After Athletic vs. Classroom Exposure.
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 3161
Participants
  COVID-19 Positive - Athletic Exposure | 24
  COVID-19 Positive - Classroom Exposure | 148
  COVID-19 Negative | 2989

11. Secondary Outcome: Number of Students With Positive COVID-19 Test After Bus vs. Classroom Exposure.
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 3161
Participants
  COVID-19 Positive - Bus Exposure | 1
  COVID-19 Positive - Classroom Exposure | 148
  COVID-19 Negative | 3012

12. Secondary Outcome: Total Number of School Days Missed Due to Symptoms After Exposure, Reported as a Mean.
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: Participants who missed school days due to symptoms after exposure.
Measure: Mean (Full Range); unit: Days
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 192
Days | 3.24737 [0 to 12]

13. Secondary Outcome: Total Number of School Days Missed Due to Isolation After Positive COVID-19 Test, Reported as a Mean.
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: Student participants who missed school days due to isolation after positive COVID-19 test.
Measure: Mean (Full Range); unit: Days
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 396
Days | 4.07888 [0 to 11]

14. Secondary Outcome: Total Number of School Days Missed Due to Quarantine After SARS-CoV-2 Exposure, Reported as a Mean.
Time Frame: up to day 7 following a known COVID-19 exposure on day 0
Population: Participants who missed school days due to quarantine after SARS-CoV-2 exposure.
Measure: Mean (Full Range); unit: Days
Arm/Group | COVID-19 Exposure Testing
Number analyzed (Participants) | 3036
Days | 0.56593 [0 to 7]

ADVERSE EVENTS:
Time Frame: Adverse Events data not collected.
Description: Adverse Events data not collected.
Arm/Group | COVID-19 Exposure Testing
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT05052580/Prot_001.pdf
  • Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT05052580/SAP_002.pdf
  • Informed Consent Form (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT05052580/ICF_000.pdf